CLINICAL TRIAL: NCT05902897
Title: Clinical Evaluation of the Braile Biomédica® Bovine Pericardium Valvular Bioprosthesis -BIOPRO TRIAL
Brief Title: Aortic or Mitral Valve Replacement With the Braile Biomédica® Bovine Pericardium Valvular Bioprosthesis
Status: Completed | Type: Observational
Sponsor: Braile Biomedica Ind. Com. e Repr. Ltda. (Industry)
Responsible Party: Sponsor
Other Study IDs: BIOPRO Trial
Record Dates: First submitted 2023-05-11; First posted 2023-06-15 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2023-06

CONDITIONS: Aortic Valve Insufficiency; Aortic Valve Regurgitation; Aortic Valve Stenosis; Aortic Valve Incompetence; Mitral Valve Insufficiency; Mitral Valve Regurgitation; Mitral Valve Stenosis; Mitral Valve Incompetence
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Valve Stenosis; Mitral Valve Insufficiency; Mitral Valve Stenosis | interventions — Replantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Braile Biomédica® Bovine Pericardium Valvular Bioprosthesis. — Heart Valve Replacement
  Other Names: Replacement for a diseased, damaged, malformed aortic or mitral heart valve

SUMMARY:
Collect data on the safety and clinical performance of the Braile Biomédica® Bovine Pericardium Valvular Bioprosthesis

DETAILED DESCRIPTION:
Multicenter, observational, retrospective, non-comparative, non-randomized study to determine the safety and clinical performance of the Bovine Pericardium Valvular Bioprosthesis in patients who required replacement of their native or bioprosthetic valve (aortic or mitral), according to ISO 14155 and ISO 5840.

ELIGIBILITY:
Inclusion Criteria:

(Group I - Aortic):

* Symptomatic patients with severe aortic insufficiency.
* Asymptomatic patients with severe aortic insufficiency and left ventricular ejection fraction (LVEF) at rest ≤ 50%.
* Patients with severe aortic insufficiency and undergoing coronary artery bypass graft surgery (CABG) or surgery of the ascending aorta or other valve.
* Asymptomatic patients with severe aortic insufficiency and resting ejection fraction > 50% with severe left ventricular (LV) dilation: left ventricular end-diastolic diameter (LVDD) > 70 mm or left ventricular ejection fraction (LVEF) > 50 mm (or LVEF > 25 mm/m2 of body surface, in patients with small body size).
* Symptomatic patients with severe high gradient aortic stenosis (mean gradient ≥ 40 mmHg or peak velocity ≥ 4.0 m/s).
* Symptomatic patients with severe low-flow, low-gradient aortic stenosis (< 40 mmHg) with reduced ejection fraction and evidence of flow reserve (contractile) excluding pseudo-severe aortic stenosis.
* Symptomatic patients with low-flow, low-gradient (< 40 mmHg) aortic stenosis with normal ejection fraction after careful confirmation of severe aortic stenosis.
* Symptomatic patients with low-flow, low-gradient aortic stenosis and reduced ejection fraction without flow reserve (contractile), particularly when the amount of calcium on computed tomography (CT) confirms severe aortic stenosis.
* Patients with symptomatic aortic stenosis at low surgical risk (STS or EuroSCORE II < 4% or logistic EuroSCORE I < 10% and no other risk factors not included in these scores, such as fragility, porcelain aorta, sequelae of thoracic radiation).
* Asymptomatic patients with severe aortic stenosis and LV systolic dysfunction (LVEF < 50%) not due to another cause.
* Asymptomatic patients with severe aortic stenosis and an abnormal exercise test showing exercise symptoms clearly related to aortic stenosis.
* Asymptomatic patients with severe aortic stenosis and an abnormal exercise test showing a decrease in blood pressure below baseline.
* Asymptomatic patients with normal ejection fraction and no exercise stress test abnormality, if the surgical risk is low and have very severe aortic stenosis defined by a peak transvalvular velocity (Vmax) > 5.5 m/s.
* Asymptomatic patients with normal ejection fraction and no exercise test abnormality, if the surgical risk is low and severe valve calcification and Vmax progression rate ≥ 0.3 m/s/year.
* Asymptomatic patients with normal ejection fraction and no exercise stress test abnormality, if surgical risk is low and B-type natriuretic peptide (BNP) marker levels are high.
* Asymptomatic patients with normal ejection fraction and no change in the exercise test, if the surgical risk is low and severe pulmonary hypertension (pulmonary artery systolic arterial pressure at rest > 60 mmHg confirmed by invasive measurement) with no other explanation.
* Patients with severe aortic stenosis undergoing CABG or surgery of the ascending aorta or other valve.
* Patients with moderate aortic stenosis undergoing CABG or surgery of the ascending aorta or other valve after decision by the Heart Team.

7.2. Inclusion Criteria (Group II - Mitral):

* Symptomatic patients with severe primary mitral insufficiency and LVEF > 30%.
* Asymptomatic patients with severe primary mitral insufficiency and LV dysfunction (LVEF > 45 mm and/or LVEF < 60%).
* Asymptomatic patients with severe primary mitral regurgitation and preserved LV function (LVEF < 45 mm and LVEF > 60%) and atrial fibrillation secondary to mitral regurgitation or pulmonary hypertension (rest systolic pulmonary pressure > 50 mmHg).
* Asymptomatic patients with severe primary mitral regurgitation and preserved LVEF (> 60%) and LVEF 40-44 mm, with leaflet failure.
* Asymptomatic patients with severe primary mitral regurgitation and preserved LVEF (> 60%) and LVEF 40-44 mm, and presence of significant LA dilation (volume index ≥ 60 mL/m2 of body surface) in sinus rhythm.
* Patients with severe primary mitral regurgitation and severe LV dysfunction (LVEF < 30% and/or LVEF > 55 mm) refractory to medical therapy.
* Patients with severe chronic secondary mitral regurgitation undergoing CABG and LVEF > 30%.
* Symptomatic patients with severe secondary mitral regurgitation, LVEF < 30%, but with the option of revascularization and evidence of myocardial viability.
* Patients with severe secondary mitral regurgitation and LVEF > 30% who remain symptomatic despite optimal clinical treatment and with low surgical risk.
* Symptomatic patients with mitral stenosis (valve area ≤ 1.5 cm2) who are not suitable for percutaneous mitral commissurotomy.

Exclusion Criteria:

* Emergency surgical valve replacement.
* Surgical replacement of the aortic root.
* Patients who did not return for follow-up examinations.
* Patients with renal impairment as determined by creatinine level ≥ 2.5 mg/dL or end-stage renal disease requiring chronic dialysis.
* Patients with stroke or transient ischemic attack within 6 months (180 days) before planned valve surgery.
* Patients with acute myocardial infarction within 30 days before planned valve surgery.
* Patients with any known life-threatening non-cardiac disease that will limit the patient's life expectancy below 1 year.
* Patients diagnosed with abnormal calcium metabolism and hyperparathyroidism.
* LVEF ≤ 20%, as validated by the diagnostic procedure before planned valve surgery.
* Echocardiographic evidence of intra-cardiac mass, thrombus or vegetation.
* Hemodynamic or respiratory instability requiring inotropic support, mechanical circulatory support, or mechanical ventilation within 30 days prior to planned valve surgery.
* Documented leukopenia (leukocytes < 3.5x10³/μL), acute anemia (Hgb < 10.0 gm/dL or 6 mmol/L) or thrombocytopenia (platelet count < 50x10³/μL) accompanied by a history of bleeding diathesis and coagulopathy.
* Patients who underwent organ transplantation.
* Pregnant or breastfeeding.
* Patients with a documented history of substance abuse (drugs or alcohol) in the last year before implantation.
* Concomitant positioning of the left ventricular assist device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing valve replacement (aortic or mitral) with Braile Biomédica® Bovine Pericardium Valvular Bioprosthesis, from 2013 to 2021.
Sampling Method: Non-Probability Sample
Enrollment: 913 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Clinical success | Until discharge from the index hospitalization (an average of 7 days is expected).
  Valve implantation without occurrences and without serious adverse events until hospital discharge.
Composite event | 01 year
  Defined as death, stroke, and/or reintervention after 1 year of follow-up.

SECONDARY OUTCOMES:
Extracorporeal circulation time AND Aortic clamping time (minutes) | during the procedure
Intensive care unit (ICU) time (days) | Until discharge from the index hospitalization (an average of 2 days is expected)
Length of in-hospital stay (days) | Until discharge from the index hospitalization (an average of 7 days is expected).
New York Heart Association (NYHA) dunctional class at 5 years post-implant compared to baseline | at discharge, 30 days, 6 months, 1 Year, 2 Years, 3 Years, 4 Years, 5 Years
  The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  Class II. Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Class III. Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV. Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
Valve related adverse events | at discharge, 30 days, 6 months, 1 Year, 2 Years, 3 Years, 4 Years, 5 Years
  structural valve deterioration, non-structural dysfunction, valve thrombosis, embolism, bleeding event, or operated valve endocarditis; death related to reintervention on the operated valve; or sudden, unexplained death
Early rates AND late linearized rates AND actuarial rates of valve-related adverse events | at discharge, 30 days, 6 months, 1 Year, 2 Years, 3 Years, 4 Years, 5 Years
  thromboembolism, valve thrombosis, all bleeds, major bleeds, paravalvular leaks, severe paravalvular leaks, endocarditis, non-structural dysfunction, structural valve deterioration (rupture and calcification)
Subject's average peak systolic gradient (mmHg) measurements at 5 years post-implant | 5 years post-implant
Subject's average mean systolic gradient (mmHg) measurements at 5 years post-implant. | 5 years post-implant
Subject's average effective orifice area measurements at 5 years post-implant | 5 years post-implant
Subject's average effective orifice area index (EOAI) measurements at 5 years post-implant | 5 years post-implant
Subject's average performance index measurements at 5 years post-implant | 5 years post-implant
Subject's average cardiac output measurements at 5 years post-implant | 5 years post-implant
Subject's amount of aortic valvular regurgitation at 5 years post-implant | 5 years post-implant

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Lucchese, Principal Investigator — Irmandade da Santa Casa de Misericordia de Porto Alegre - ISCMPA
Locations (3):
- Brazil (3):
  - Hospital Ana Nery - HAN/SESAB, Salvador, Estado de Bahia
  - Irmandade da Santa Casa de Misericordia de Porto Alegre - ISCMPA, Porto Alegre, Rio Grande do Sul
  - InCor - Instituto do Coração do Hospital das Clínicas da FMUSP, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No